CLINICAL TRIAL: NCT02178865
Title: Evaluation of the Accuracy of Predicting Normal or Carrier Status in Euploid Embryos Produced by Patients With Balanced Translocations
Brief Title: Predicting Normal vs. Carrier Status in Euploid Embryos of Translocation Carriers
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2014-01
Record Dates: First submitted 2014-06-26; First posted 2014-07-01 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Balanced Chromosomal Translocation
Keywords: translocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — buccal swabs and whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- translocation carrier: balanced translocation carriers who have undergone IVF

SUMMARY:
The purpose of this study is to assess the accuracy of predicting the normal or carrier status of human embryos resulting from in vitro-fertilization (IVF) from patients carrying a balanced translocation.

DETAILED DESCRIPTION:
This study aims to evaluate the validity of using informative SNPs to distinguish balanced from normal embryos. This will involve acquiring material from families to set phase for informative SNPs, evaluation of existing and new embryo SNP array data, and follow up analysis of children born after applying the procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients with balanced translocations who have undergone IVF

Exclusion Criteria:

* those who do not wish to know their child(s) karyotype

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with balanced translocations
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Proportion of correct predictions of normal vs. balanced ploidy status as compared to conventional karyotype | up to 12 months once pregnant

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, HCLD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No